CLINICAL TRIAL: NCT07002515
Title: THE EFFECT OF HEALTH EDUCATION ON DIGITAL GAME ADDICTION AND HEALTH PROMOTION BEHAVIOR IN ADOLESCENTS
Acronym: Digital Addict
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Serpil Özdemir, PhD, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-29
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Internet Addiction Disorder; Health Promotion
Keywords: Digital Technology; Health Promotion; Internet Addiction Disorder; Health Education; Adolescent
MeSH Terms: conditions — Internet Addiction Disorder; Health Education

STUDY DESIGN:
Intervention Model Description: A four-arm randomized controlled study using the Solomon design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Group 1 (Experimental): contains 40 adolescents
  Interventions: Other: Health education
- Intervention Group 2 (Experimental): contains 40 adolescents
  Interventions: Other: Health education
- Control Group 1 (No Intervention): contains 40 adolescents
- Control Group 2 (No Intervention): contains 40 adolescents

INTERVENTIONS:
Other: Health education — Randomized controlled studies that explain behavior change as a process through health education aimed at promoting healthy behaviors in individuals with digital game addiction.
  Other Names: Prevention of digital game addiction
  Arms: Intervention Group 1; Intervention Group 2

SUMMARY:
Nowadays, among adolescents who are frequently exposed to digital technologies, problematic behaviors resulting from misuse such as problematic internet use, video game addiction, and online gaming disorder are commonly observed (Young, 2017). In the literature, the prevalence of digital game addiction among adolescents has been reported to range between 0.7% and 15.6% (Arifin et al., 2022; Karadağ & Noyan, 2023; Miezaha et al., 2020; Yudes et al., 2021). Promoting health-enhancing behaviors plays a key role in combating digital game addiction in adolescent health (Daysal & Yılmazel, 2020). Previous studies have found that adolescents generally exhibit a moderate level of health-promoting behaviors (Özdemir & Bülbül, 2023). When behaviors such as regular sleep, stress management, exercise, and adequate and balanced nutrition are adopted by adolescents with the aim of improving health, the need for technology tends to decrease (Bebiş et al., 2015; Özcan et al., 2023; Hysing et al., 2021).

When the existing literature is reviewed, it appears that there is a lack of randomized controlled trials that explain behavior change as a process through health education aimed at promoting healthy behaviors among individuals affected by digital game addiction, which is considered a significant problem in adolescents (Shinde et al., 2020; Yang, 2020). In this context, the aim of this study is to determine the effect of health education provided to adolescents on digital game addiction and health-promoting behaviors.

The population of the study consisted of 5th, 6th, 7th, and 8th grade students (n = 825) enrolled at Etimesgut 15 July Martyrs Secondary School located in the city center of Ankara. When the study was completed with 136 participants, a post hoc power analysis indicated that with an effect size of f = 0.25, the study achieved 80% power and 95% confidence (1-α) based on a four-group experimental design with repeated measures ANOVA, with a minimum of 34 participants per group (Cohen, 1992). Considering potential participant loss, the sample size was increased by 15%, and the study was initiated with 160 participants, allocating 40 to each group.

The study will begin after obtaining permission from the Ankara Provincial Directorate of National Education and approval from the Ethics Committee. Following the identification of voluntary adolescents who meet the inclusion criteria, information about the study will be provided to both the adolescents and their parents, and written informed consent will be obtained. In this randomized controlled study based on the Solomon four-group design, participants will be assigned to groups using the block randomization method (Group 1: Intervention Group 1, Group 2: Intervention Group 2, Group 3: Control Group 1, Group 4: Control Group 2). Research data will be collected through a pretest administered to Group 1 (intervention 1) and Group 3 (control 1) immediately after randomization and prior to training, and a post-test administered to all groups at the end of the third month following the completion of the four training sessions.

The intervention groups will receive a standardized health education program delivered over four sessions spanning three months. The timing of the training sessions will be coordinated with the school administration to fit within the school schedule. The data collection tools used in the study include the Descriptive Information Form (20 items), the Digital Game Addiction Scale for Children (24 items), and the Adolescent Health Promotion Scale (40 items).

If the data do not follow a normal distribution, non-parametric methods will be used, and analyses will be conducted using the Walrus package in the JAMOVI software. For analyzing the relationships between scales, Pearson or Spearman correlation coefficients will be used depending on the normality of the data. For categorical data, if the expected frequency is greater than 25, Pearson's chi-square test will be applied; if it is between 5 and 25, Yates' correction will be used; and if it is less than 5, Fisher's exact test will be employed. For the analysis of numerical demographic data, one-way ANOVA will be used if the data are normally distributed, and the Kruskal-Wallis test will be used if not. IBM SPSS Statistics version 23 will be used for statistical evaluations. A significance level of p < 0.05 will be considered statistically significant in this study.

DETAILED DESCRIPTION:
PURPOSE AND SIGNIFICANCE OF THE STUDY

Today, the use of digital technologies is highly prevalent in all societies where internet access is widespread and easily accessible, particularly in developed countries (Akgül et al., 2021; Li et al., 2021; Yang, 2020). Among adolescents who are frequently exposed to digital technologies, problematic behaviors resulting from misuse-such as problematic internet use, video game addiction, and online gaming addiction-are commonly observed (Young, 2017). Another significant issue under the umbrella of digital technology addiction is digital game addiction. Digital game addiction is defined as a behavioral addiction that is frequently encountered among adolescents (Daysal & Yılmazel, 2020; Tunç, 2023). According to the literature, the prevalence of digital game addiction among adolescents ranges from 0.7% to 15.6% (Arifin et al., 2022; Karadağ & Noyan, 2023; Miezaha et al., 2020; Yudes et al., 2021). Promoting health-enhancing behaviors plays a key role in combating digital game addiction in adolescent health (Daysal & Yılmazel, 2020). To adopt health-promoting behaviors, adolescents need to establish self-control and aim to adopt positive health behaviors. Studies have shown that adolescents' levels of health-promoting behavior are at a moderate level (Özdemir & Bülbül, 2023). This indicates that adolescents need to be further supported in developing and maintaining positive health behaviors (Özdemir & Bülbül, 2023). When adolescents are encouraged to adopt behaviors that promote health-such as regular sleep, stress management, exercise, and a balanced and adequate diet-their dependence on and need for technology can be diminished (Bebiş et al., 2015; Özcan et al., 2023; Hysing et al., 2021). Research conducted around the world also identifies the prevention of digital game addiction among adolescents as a top priority and a significant public health issue (Li et al., 2021; Miezaha et al., 2020).

Upon examining the existing studies, it is evaluated that there is an insufficient number of randomized controlled studies that explain the process of behavioral change through health education aimed at instilling healthy behaviors in adolescents, for whom digital game addiction is considered a major issue (Shinde et al., 2020; Yang, 2020). In this context, the aim of this study is to determine the effect of health education provided to adolescents on digital game addiction and health-promoting behaviors.

Design, Setting, and Characteristics of the Study The study is planned to be conducted as a four-group randomized controlled trial using the Solomon design between February 2025 and June 2025 at Etimesgut 15 Temmuz Şehitleri Middle School, which is affiliated with the Ankara Provincial Directorate of National Education.

Population and Sample of the Study The population of the study consisted of 5th, 6th, 7th, and 8th grade students (n = 825) enrolled at Etimesgut 15 Temmuz Şehitleri Middle School, located in Ankara city center. A post hoc power analysis indicated that the study would require a minimum of 34 participants per group-136 participants in total-to achieve 80% power at a 95% confidence level (1-α), assuming an effect size of f = 0.25 and based on repeated measures ANOVA for a four-group experimental design model (Cohen, 1992). Considering potential dropouts, the sample size was increased by 15%, and the study was initiated with a total of 160 participants, with 40 individuals in each group.

Inclusion Criteria

Currently enrolled and attending education at the school where the study is conducted

Living with parents

Owning a technical device such as a mobile phone, tablet, computer, or gaming console, and actively playing digital games

Having voluntary informed consent from both the parent and the adolescent

Exclusion Criteria Having psychiatric or educational difficulties such as attention deficit and hyperactivity disorder (ADHD), specific learning disabilities, intellectual disability, or speech and language impairments

Withdrawal Criteria Voluntarily leaving the study Missing at least one session of the health education intervention Data Collection Tools

1. Introductory Information Forms The research data will be collected using Introductory Information Forms developed by the researchers based on the relevant literature.

   Form I includes questions about gender, year of birth, parents' education and employment status, duration and purpose of internet use, types of digital games played, and experiences of peer bullying.

   Form II includes questions about the duration and frequency of digital gameplay, and the effectiveness of the provided education.
2. Digital Game Addiction Scale for Children (DGASC) Developed by Hazar and Hazar (2017) to assess digital game addiction levels in children aged 10-14. The scale is a 5-point Likert-type instrument consisting of 24 items and 4 subscales.

   Each item is rated as follows:

   "1 = Strongly Disagree", "2 = Disagree", "3 = Neutral", "4 = Agree", "5 = Strongly Agree". The lowest possible score is 24, and the highest is 120.

   The score interpretation is as follows:

   1-24: Normal group

   25-48: Low-risk group

   49-72: Risk group

   73-96: Addicted group

   97-120: Highly addicted group

   The subscales include:

   Excessive Focus on and Conflict Over Playing Digital Games

   Tolerance Development and Value Attribution to Game Time

   Postponement of Individual and Social Responsibilities

   Psychological and Physiological Withdrawal Symptoms and Immersion in Games

   The Cronbach's alpha coefficient for the entire scale is 0.90, and for the subscales, they are 0.78, 0.81, 0.76, and 0.67 respectively. There are no reverse-coded items.
3. Adolescent Health Promotion Scale (AHPS) The AHPS was developed by Mei-Yen Chen et al. in 2003. Its Turkish validity and reliability were established by Ortabağ et al. (2011) and Bayık Temel et al. (2011).

   Both studies concluded that the scale is valid and reliable for use in Turkish society.

   The Cronbach's alpha reliability of the scale is reported as 0.86.

   The scale consists of 40 items and six subscales:

   Nutrition (6 items)

   Interpersonal Support (7 items)

   Health Responsibility (8 items)

   Self-Actualization (8 items)

   Exercise (4 items)

   Stress Management (6 items)

   Items are rated using a 5-point Likert scale:

   "1 = Never", "2 = Sometimes", "3 = Usually", "4 = Often", "5 = Always". Each subscale score is obtained by summing its items; the total score is the sum of all subscale scores. The total score ranges from 40 to 200.

   Health Education In this study, a health education intervention will be delivered using a slide presentation and printed/digital brochures.

   The content was developed based on relevant literature to meet participants' informational needs, raise awareness, foster safe and limited digital gameplay habits, and help sustain these behaviors.

   Additionally, educational materials were informed by national resources such as:

   "Conscious, Safe, and Effective Use of Information Technologies"

   "Parental Guide for Protecting Children from Digital Risks"

   "Before Technology Turns into a Monster!" (Turkey Addiction Prevention Training Program)

   "Technology Addiction" brochures

   Topics covered in the health education slide presentation include:

   Prevalence of digital technology addiction

   Signs of digital addiction and coping strategies

   Ways to overcome digital game addiction

   Importance of managing and sustaining this process in a healthy way

   Importance of protecting and promoting health

   Importance of balanced nutrition, physical activity, and healthy sleep patterns

   Importance of maintaining health-promoting behaviors

   Concept of digital citizenship

   Importance of being a conscious digital literate

   Safe and effective use of information and communication technologies

   Recommended websites

   The health education brochure includes:

   Signs and risk factors of digital game addiction

   Strategies to overcome addiction, including alternative sports and social hobbies

   Physical activity, balanced nutrition, and sleep hygiene

   Promotion of the "Safe Internet Center" website

   The brochure served as a complementary and reminder tool supporting the health education.

   Implementation of the Study The study will begin after receiving approval from the Ankara Provincial Directorate of National Education and an Ethics Committee.

   Voluntary adolescents who meet the inclusion criteria will be identified. Before the intervention, both adolescents and their parents will be informed about the study and written consent will be obtained.

   Participants will be randomly assigned to one of four groups using block randomization within the Solomon four-group randomized controlled trial design:

   Group 1: Intervention Group 1

   Group 2: Intervention Group 2

   Group 3: Control Group 1

   Group 4: Control Group 2

   Data will be collected at two time points:

   A pre-test for Group 1 (Intervention 1) and Group 3 (Control 1) before the first session

   A post-test for all four groups at the end of month 3 (after completing four health education sessions)

   The intervention groups will receive a standardized health education program spanning three months, consisting of four sessions.

   Session times will be scheduled in cooperation with the school administration according to the academic timetable.

   Pre-test tools include:

   Introductory Information Form (20 items)

   Digital Game Addiction Scale for Children (24 items, with four subscales: Excessive Focus and Conflict, Tolerance and Value Attribution, Postponement of Responsibilities, Psychological-Physiological Withdrawal)

   Adolescent Health Promotion Scale (40 items, with six subscales: Nutrition, Interpersonal Support, Health Responsibility, Self-Actualization, Exercise, and Stress Management)

   Written permissions have been obtained from the primary authors of the scales used in the study.

   Data Analysis If data are normally distributed, generalized linear models will be used to compare digital game addiction and health promotion scores across groups and over time.

   If not normally distributed, non-parametric methods will be applied, and analysis will be conducted using the JAMOVI software with the Walrus package.

   Correlations between scales will be examined using Pearson or Spearman correlation coefficients depending on the distribution.

   For all categorical data, depending on the minimum expected frequency:

   Pearson's chi-square test will be used if all values exceed 25

   Yates' correction if values are between 5 and 25

   Fisher's exact test if values are below 5

   For quantitative demographic data:

   One-way ANOVA will be used if data are normally distributed

   Kruskal-Wallis test if not

   All statistical analyses will be performed using IBM SPSS Statistics version 23.

   A p-value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and continuing education at the center where the study is conducted
* Living with their parents
* Owning a technical device such as a mobile phone/tablet/computer/game console and playing digital games
* Having voluntary consent from both the adolescent and their parents

Exclusion Criteria:

* Having psychiatric or educational difficulties such as attention deficit and hyperactivity disorder, specific learning disabilities, intellectual disabilities, language and speech impairments, etc.
* Voluntarily withdrawing from the study
* Not attending at least one session of the health education program

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Children's Digital Game Addiction Scale | 3 months
  It was developed by Hazar and Hazar (2017) to determine the levels of digital game addiction in children aged 10-14. The scale, prepared as a 5-point Likert type, consists of 4 sub-factors and 24 items. Each item on the scale is coded as "1 = Strongly Disagree," "2 = Disagree," "3 = Neutral," "4 = Agree," and "5 = Strongly Agree." The lowest possible score on the scale is 24, and the highest is 120. The scoring classification is as follows: "1-24: Normal group, 25-48: Low-risk group, 49-72: Risk group, 73-96: Addicted group, 97-120: Highly addicted group." The sub-dimensions of the scale are: "Excessive Focus and Conflict Related to Digital Gaming," "Tolerance Development in Game Time and Value Assigned to the Game," "Postponement of Individual and Social Tasks/Homework," and "Psychological-Physiological Reflection of Withdrawal and Immersion in the Game." The Cronbach's alpha for the entire scale is 0.90, and for the sub-factors, it is 0.78, 0.81, 0.76, and 0.67, respectively.
Adolescent Health Promotion Scale | 3 months
  The Adolescent Health Promotion Scale (AHPS) was developed by Mei-Yen Chen and colleagues in 2003. Its Turkish validity and reliability studies were conducted by Ortabağ et al. (2011) and Bayık Temel et al. (2011), and both studies indicated that the scale is valid and reliable for use in the Turkish population. The scale's Cronbach's alpha reliability coefficient is reported as 0.86.
  The Adolescent Health Promotion Scale consists of 40 items. Its subscales are nutrition (6 items), interpersonal support (7 items), health responsibility (8 items), self-actualization (8 items), exercise (4 items), and stress management (6 items). The items are rated on a 5-point Likert scale as follows: "1 = never, 2 = sometimes, 3 = usually, 4 = often, 5 = always."
  Scores for each subscale are obtained by summing the item scores within that subscale, and the total scale score is obtained by summing all subscale scores. The possible total score ranges from 40 to 200.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi Gulhane Hemsirelik Fakultesi, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen MY, Wang EK, Yang RJ, Liou YM. Adolescent health promotion scale: development and psychometric testing. Public Health Nurs. 2003 Mar-Apr;20(2):104-10. doi: 10.1046/j.1525-1446.2003.20204.x. PMID 12588427
- [Background] Ortabag T, Ozdemir S, Bakir B, Tosun N. Health promotion and risk behaviors among adolescents in Turkey. J Sch Nurs. 2011 Aug;27(4):304-15. doi: 10.1177/1059840511408322. Epub 2011 May 6. PMID 21551314
- [Background] Hazar, Z., ve Hazar, M. (2017). Çocuklar İçin Dijital Oyun Bağımlılığı Ölçeği. Journal of Human Sciences, 14(1), 203-216. Doi:10.14687/jhs.v14i1.4387
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Shinde S, Weiss HA, Khandeparkar P, Pereira B, Sharma A, Gupta R, Ross DA, Patton G, Patel V. A multicomponent secondary school health promotion intervention and adolescent health: An extension of the SEHER cluster randomised controlled trial in Bihar, India. PLoS Med. 2020 Feb 11;17(2):e1003021. doi: 10.1371/journal.pmed.1003021. eCollection 2020 Feb. PMID 32045409
- [Background] Hysing M, Askeland KG, La Greca AM, Solberg ME, Breivik K, Sivertsen B. Bullying Involvement in Adolescence: Implications for Sleep, Mental Health, and Academic Outcomes. J Interpers Violence. 2021 Sep;36(17-18):NP8992-NP9014. doi: 10.1177/0886260519853409. Epub 2019 Jun 10. PMID 31179829
- [Background] Özcan, M., Polat, T.ve Alkan-Polat, B. (2023). Adölesanlarda E-Sağlık Okuryazarlığının Sağlığı Geliştirme Davranışına Etkisi, Gümüşhane Üniversitesi Sağlık Bilimleri Dergisi, 12(3), 1060- 1071
- [Background] Bebiş, H., Akpunar, A., Özdemir, S. ve Kılıç, S.(2015). Bir Ortaöğretim Okulundaki Adölesanların Sağlığı Geliştirme Davranışlarının İncelenmesi. Gülhane Tıp Dergisi, 57, 129-135.
- [Background] Özdemir, S. ve Bülbül, F.(2023) Adölesanlarda Sağlığı Geliştirme ve Yaşamda Anlam Arasındaki İlişki. Hacettepe Üniversitesi Hemşirelik Fakültesi Dergisi, 10(1):1- 8. DOI: 10.31125/hunhemsire.1272589
- [Background] Yudes C, Rey L, Extremera N. The Moderating Effect of Emotional Intelligence on Problematic Internet Use and Cyberbullying Perpetration Among Adolescents: Gender Differences. Psychol Rep. 2022 Dec;125(6):2902-2921. doi: 10.1177/00332941211031792. Epub 2021 Jul 9. PMID 34240633
- [Background] Miezah, D., Batchelor, J., Megreya, A.M., Richard Y. ve Moustafa A.A. (2020). Video/Computer Game Addiction among University Students in Ghana: Prevalence, Correlates and Effects of Some Demographic Factors. Psychiatry and Clinical Psychopharmacology.30(1):17-23. Doi:10.5455/PCP.20200320092210.
- [Background] Karadağ, Y. E. ve Noyan, C. O. (2023) Teknoloji Bağımlılığını Önlemeye Yönelik Psikoeğitim Programının 8. Sınıf Öğrencileri Üzerindeki Etkisi. Bağımlılık Dergisi, 24(1), 43-52. Doi: 10.51982/bagimli.1090570.
- [Background] Arifin, R., Wedhatami, B., Alkadri, R. ve Daniel, N. (2022). The internet gang of violence: Trend of cyberbullying on the internet. AIP Conference Proceedings, 2573, 040012-1- 040012-5.
- [Background] Tunç,C.(2023).Lise Öğrencilerinde Dijital Oyun Bağımlılığı ve Siber Zorbalık. Yayınlanmamış Yüksek Lisans Tezi,Van Yüzüncüyıl Eğitim Bilimleri Enstitüsü, Van.
- [Background] Daysal, B., ve Yılmazel, G. (2020). Halk Sağlığı Gözüyle Akıllı Telefon Bağımlılığı ve Ergenlik. Turkish Journal of Family Medicine and Primary Care, 14(2), 316-322. Doi: 10.21763/tjfmpc.730254.
- [Background] Young, K. S. (2017). Assessment Issues with Internet-Addicted Children and Adolescents. In Young, K.S. and de Abreu, C.N., Eds., Internet Addiction in Children and Adolescents: Risk Factors, Assessment, and Treatment. Springer Publishing Company, New York, 143-160. Doi: 10.1891/9780826133731.0008
- [Background] Yang SY. Effects of Self-efficacy and Self-control on Internet Addiction in Middle School Students: A Social Cognitive Theory-Driven Focus on the Mediating Influence of Social Support. Child Health Nurs Res. 2020 Jul;26(3):357-365. doi: 10.4094/chnr.2020.26.3.357. Epub 2020 Jul 31. PMID 35004479
- [Background] Li S, Ren P, Chiu MM, Wang C, Lei H. The Relationship Between Self-Control and Internet Addiction Among Students: A Meta-Analysis. Front Psychol. 2021 Nov 24;12:735755. doi: 10.3389/fpsyg.2021.735755. eCollection 2021. PMID 34899477